CLINICAL TRIAL: NCT04117126
Title: Efficacy of Prompted Voiding Therapy for Reverse the Urinary Incontinence Status in Elderly Patients Hospitalized in a Functional Recovery Ward.
Brief Title: Efficacy of Prompted Voiding Therapy in Elderly Hospitalized.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guadarrama Hospital (Other)
Responsible Party: Principal Investigator, Laura Martín Losada, Registered Nurse, Doctoral student., Guadarrama Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7.0
Record Dates: First submitted 2019-08-17; First posted 2019-10-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Urinary Incontinence
Keywords: aged; Therapeutics; hospitalization; nursing care; rehabilitation; prompted voiding
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- urinary incontinence (Experimental): Recruitment, 3-day voiding record, initiate a individualized prompted voiding schedule based on the client's toileting needs until discharge, 1, 3 and 6 month follow-up post-discharge.
  Interventions: Behavioral: Prompted voiding

INTERVENTIONS:
Behavioral: Prompted voiding — Monitoring: This involves asking the incontinent individual, at regular intervals, if he or she needs to use the toilet. The care provider may look for behaviours that the client needs to be toileted (e.g., restlessness, agitation, disrobing), and take the client to the toilet at regular intervals specific to their schedule, rather than routinely every two hours.
  Prompting: This process includes prompting the person to use the toilet at regular intervals, and encourages the maintenance of bladder control between prompted voiding sessions.
  Praising: This important step is the positive reinforcement of dryness and appropriate toileting, and is the response from the care provider to the individual's success with maintaining bladder control.

SUMMARY:
This study evaluates effectiveness to apply prompted voiding in urinary incontinence and dependence patients admitted at functional recovery ward in a mid-stay hospital. This behavioural therapy is recommended in Best Practice Guidelines, and it has good results in elderly living in the community or in nursing home but yet it has not shown his benefits in hospitalized elderly patients for a long time.

DETAILED DESCRIPTION:
The increased level of chronic diseases, greater chances of survival and older people hospitalized, place the Urinary Incontinence (UI) problem in a priority position both in hospital and community care. Guadarrama (Public Madrid Health Service) is a medium-stay Hospital. It makes treatment to recover from acute disease and UI has 80% prevalence at admitted patients.

Main objective:To assess the efficacy of Prompted Voiding (PV) therapy for reverse of UI status in elderly patients hospitalized in a Functional Recovery Ward. (FRW) Methods: Experimental research pre/post-Intervention, with 5 repeated measures data: baseline (preintervention); at discharge, at one, three and six months after discharge (post-intervention). Sample size is 212 admitted patients in the FRW with UI. Prompted voiding intervention will be applied by nursing team following the procedure hospital approved and it will be individualized to each patient.

Main Outcome: urinary continence (YES/NO), others outcomes: amount and frequency of urine loss, type of incontinence pads; follow-up: urinary continence at one, three, and six months after discharge.

Applicability: Incorporating Prompted Voiding Therapy in UI patients care, encouraging global care, relevant implications for reduce the morbidity, improvement the quality of life, decrease health costs.

ELIGIBILITY:
Inclusion Criteria:

* onset of Urinary Incontinence less than 1 year (information extracted from the Patient's Medical History, or provided by the patient or family caregiver)
* sign the informed consent.

Exclusion Criteria:

* patient with indwelling urinary catheters at admission
* irreversible urinary incontinence by disease itself
* moderate-severe cognitive impairment (Pfeiffer's questionnaire > 4)
* patients with indication of water restriction.
* patients who do not collaborate in Prompted Voiding therapy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 158 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Change of Urinary Incontinence status after prompted voiding program (PVP) | at admission, at discharge (about 30 to 60 days), 1 , 3 and 6 month post discharge
  To value the efficacy of prompted voiding therapy to recovery urinary continence in elderly hospitalized at functional recovery ward. Data wil be collected from nursing assessment at admission, at discharge and telephone call.
Improve urinary incontinence episodes/symptoms after prompted voiding program. | at admission, each 15 days along admission, at discharge (about 30 to 60 days).
  To value the efficacy of prompted voiding therapy to improve urinary incontinence episodes/symptoms (episodes frequency, volume loss, type pad used) in elderly hospitalized at functional recovery ward. It Will be measure with assistance nurse record.

SECONDARY OUTCOMES:
Change of Urinary Incontinence status after PVP in admitted patients with Stress Urinary Incontinence | at admission, at discharge.(about 30 to 60 days)
  Assessment will be with IU4 questionnaire and NANDA diagnosis. Data will be collected from nursing assessment at admission and nursing assesment at discharge records.
Change of Urinary Incontinence status after PVP in admitted patients with Emergency Urinary Incontinence | at admission, at discharge.(about 30 to 60 days)
  Assessment will be with IU4 questionnaire and NANDA diagnosis. Data will be collected from nursing assessment at admission and nursing assesment at discharge records.
Change of Urinary Incontinence status after PVP in admitted patients with Mixed Urinary Incontinence | at admission, at discharge.(about 30 to 60 days)
  Assessment will be with IU4 questionnaire and NANDA diagnosis. Data will be collected from nursing assessment at admission and nursing assesment at discharge records.
Change of Urinary Incontinence status after PVP in admitted patients with Functional Urinary Incontinence | at admission, at discharge.(about 30 to 60 days)
  Assessment will be with IU4 questionnaire and NANDA diagnosis. Data will be collected from nursing assessment at admission and nursing assesment at discharge records.
Change from Urinary Incontinence status after PVP in admitted patients with Reflects Urinary Incontinence | at admission, at discharge.(about 30 to 60 days)
  Assessment will be with IU4 questionnaire and NANDA diagnosis. Data will be collected from nursing assessment at admission and nursing assesment at discharge records.
Change of Urinary Incontinence status after PVP in admitted patients with Total Urinary Incontinence | at admission, at discharge.(about 30 to 60 days)
  Assessment will be with IU4 questionnaire and NANDA diagnosis. Data will be collected from nursing assessment at admission and nursing assesment at discharge records.
Urinary Incontinence (UI) status reached related with aged. | at admission, at discharge (about 30 to 60 days)
  To Identify promoting/difficulty continence factors. Data will be collected from clinical history records.
Urinary Incontinence (UI) status reached related with cognitive ability. | at admission, at discharge (about 30 to 60 days)
  To Identify promoting/difficulty continence factors. Data will be collected from clinical history records. Cognitive impairments will be measure with Pfeiffer test.
Urinary Incontinence (UI) status reached related with Functional ability. | at admission, at discharge (about 30 to 60 days)
  To Identify promoting/difficulty continence factors. Data will be collected from clinical history records. Functional ability will be measure with Barthel Scale.
Urinary Incontinence (UI) status reached related with risk diseases presence. | at admission, at discharge (about 30 to 60 days)
  To Identify promoting/difficulty continence factors. Data will be collected from clinical history records. Risk diseases: Diabetes Mellitus, Parkinson Disease, Heart Failure, Obesity, Urinary Tract infection, Nervous System Diseases, Stroke, Abdomen and pelvis surgery.
Urinary Incontinence (UI) status reached related with risk drugs. | at admission, at discharge (about 30 to 60 days)
  To Identify promoting/difficulty continence factors. Data will be collected from clinical history records and drug prescriptions. Risk drugs: Diuretics; sedatives; hypnotics; anticholinergics; amitriptyline; opioid analgesics, cholinesterase inhibitors.
Urinary Incontinence (UI) status reached related with overweigth. | at admission, at discharge (about 30 to 60 days)
  To Identify promoting/difficulty continence factors. Data will be collected from clinical history records. Body Mass Index greater than or equal to 25
Urinary Incontinence (UI) status reached related with caregiver presence. | at admission, at discharge (about 30 to 60 days)
  To Identify promoting/difficulty continence factors. Data will be collected from clinical history records.
Urinary Incontinence (UI) status reached related to diagnosis of admission | at admission, at discharge (about 30 to 60 days)
  To Identify promoting/difficulty continence factors. Data will be collected from clinical history records. 3 groups will be assigned: Femoral Fractures, stroke, functional disability.
Urinary Incontinence (UI) status reached related to risk of Skin Ulcer | at admission, at discharge (about 30 to 60 days)
  Data will be collected from clinical history records. It will be valuated with Norton Scale.
Urinary Incontinence (UI) status reached related to fall risk. | at admission, at discharge (about 30 to 60 days)
  Data will be collected from clinical history records. It will be valuated with Sytratify Scale.
Urinary Incontinence (UI) status reached related to days of hospitalization. | at admission, at discharge (about 30 to 60 days)
  To Identify promoting/difficulty continence factors. Data will be collected from clinical history records.
Urinary Incontinence (UI) status reached related with time of UI. | at admission, at discharge (about 30 to 60 days)
  To Identify promoting/difficulty continence factors. Data will be collected from clinical history records.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Martin Losada, Principal Investigator — Hospital Guadarrama
Locations (1):
- Laura Martín Losada, Guadarrama, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jansen APD, Muntinga ME, Bosmans JE, Berghmans B, Dekker J, Hugtenburgh J, Nijpels G, van Houten P, Laurant MGH, van der Vaart HCH. Cost-effectiveness of a nurse-led intervention to optimise implementation of guideline-concordant continence care: Study protocol of the COCON study. BMC Nurs. 2017 Feb 22;16:10. doi: 10.1186/s12912-017-0204-8. eCollection 2017. PMID 28239296
- [Background] Thuroff JW, Abrams P, Andersson KE, Artibani W, Chapple CR, Drake MJ, Hampel C, Neisius A, Schroder A, Tubaro A; European Association of Urology. [EAU Guidelines on Urinary Incontinence]. Actas Urol Esp. 2011 Jul-Aug;35(7):373-88. doi: 10.1016/j.acuro.2011.03.012. Epub 2011 May 19. Spanish. PMID 21600674
- [Background] Promoting Continence Using Prompted Voiding Guideline. [Internet] RNAO, 2011. Available in https://rnao.ca/bpg/guidelines/promoting-continence-using-prompted-voiding
- [Background] Terzoni S, Montanari E, Mora C, Destrebecq A. Urinary incontinence in adults: nurses' beliefs, education and role in continence promotion. A narrative review. Arch Ital Urol Androl. 2011 Dec;83(4):213-6. PMID 22670322
- [Background] Baztan JJ, Arias E, Gonzalez N, Rodriguez de Prada MI. New-onset urinary incontinence and rehabilitation outcomes in frail older patients. Age Ageing. 2005 Mar;34(2):172-5. doi: 10.1093/ageing/afi001. No abstract available. PMID 15713862
- [Background] Riemsma R, Hagen S, Kirschner-Hermanns R, Norton C, Wijk H, Andersson KE, Chapple C, Spinks J, Wagg A, Hutt E, Misso K, Deshpande S, Kleijnen J, Milsom I. Can incontinence be cured? A systematic review of cure rates. BMC Med. 2017 Mar 24;15(1):63. doi: 10.1186/s12916-017-0828-2. PMID 28335792
- [Background] Holtzer-Goor KM, Gaultney JG, van Houten P, Wagg AS, Huygens SA, Nielen MM, Albers-Heitner CP, Redekop WK, Rutten-van Molken MP, Al MJ. Cost-Effectiveness of Including a Nurse Specialist in the Treatment of Urinary Incontinence in Primary Care in the Netherlands. PLoS One. 2015 Oct 1;10(10):e0138225. doi: 10.1371/journal.pone.0138225. eCollection 2015. PMID 26426124
- [Background] Lai CKY, Wan X. Using Prompted Voiding to Manage Urinary Incontinence in Nursing Homes: Can It Be Sustained? J Am Med Dir Assoc. 2017 Jun 1;18(6):509-514. doi: 10.1016/j.jamda.2016.12.084. Epub 2017 Feb 22. PMID 28236604
- [Background] Gibson JM, Thomas LH, Harrison JJ, Watkins CL; ICONS Project Team and the ICONS Patient, Public and Carer Involvement Groups. Stroke survivors' and carers' experiences of a systematic voiding programme to treat urinary incontinence after stroke. J Clin Nurs. 2018 May;27(9-10):2041-2051. doi: 10.1111/jocn.14346. PMID 29517816
- [Background] Suzuki M, Iguchi Y, Igawa Y, Yoshida M, Sanada H, Miyazaki H, Homma Y. Ultrasound-assisted prompted voiding for management of urinary incontinence of nursing home residents: Efficacy and feasibility. Int J Urol. 2016 Sep;23(9):786-90. doi: 10.1111/iju.13156. Epub 2016 Jul 11. PMID 27399836
- [Background] Thomas LH, French B, Burton CR, Sutton C, Forshaw D, Dickinson H, Leathley MJ, Britt D, Roe B, Cheater FM, Booth J, Watkins CL; ICONS Project Team; ICONS Patient, Public and Carer Involvement Groups. Evaluating a systematic voiding programme for patients with urinary incontinence after stroke in secondary care using soft systems analysis and Normalisation Process Theory: findings from the ICONS case study phase. Int J Nurs Stud. 2014 Oct;51(10):1308-20. doi: 10.1016/j.ijnurstu.2014.02.009. Epub 2014 Feb 20. PMID 24656435
- [Background] Holroyd-Leduc JM, Straus SE. Management of urinary incontinence in women: scientific review. JAMA. 2004 Feb 25;291(8):986-95. doi: 10.1001/jama.291.8.986. PMID 14982915
- [Background] Franken MG, Corro Ramos I, Los J, Al MJ. The increasing importance of a continence nurse specialist to improve outcomes and save costs of urinary incontinence care: an analysis of future policy scenarios. BMC Fam Pract. 2018 Feb 17;19(1):31. doi: 10.1186/s12875-018-0714-9. PMID 29454331
- [Background] Eustice S, Roe B, Paterson J. Prompted voiding for the management of urinary incontinence in adults. Cochrane Database Syst Rev. 2000;2000(2):CD002113. doi: 10.1002/14651858.CD002113. PMID 10796861
- [Background] Morilla JC, Iglesias J, Izquierdo JM, Martín MJ, Martín MC, Rodríguez C. et al. Guía de atención enfermera a pacientes con incontinencia urinaria. Asociación Andaluza de Enfermería Comunitaria, 2007.
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] Barentsen JA, Visser E, Hofstetter H, Maris AM, Dekker JH, de Bock GH. Severity, not type, is the main predictor of decreased quality of life in elderly women with urinary incontinence: a population-based study as part of a randomized controlled trial in primary care. Health Qual Life Outcomes. 2012 Dec 18;10:153. doi: 10.1186/1477-7525-10-153. PMID 23249635
- [Background] García M. Análisis descriptivo del gasto sanitario español: evolución, desglose, comparativa internacional y relación con la renta. [Internet] Instituto de Estudios Fiscales. I.S.S.N.: 1578-0252 Available in http://www.ief.es/documentos/recursos/publicaciones/papeles_trabajo/2006_24.pdf
- [Background] Miner PB Jr. Economic and personal impact of fecal and urinary incontinence. Gastroenterology. 2004 Jan;126(1 Suppl 1):S8-13. doi: 10.1053/j.gastro.2003.10.056. PMID 14978633
- [Background] Baena V, Blasco P, Cozar-Olmo JM, Díez-Itza I, Espuña M, Hidalgo A. Libro Blanco de la Carga Socioeconómica de la Incontinencia Urinaria en España, 2017.
- [Background] Martinez Agullo E, Ruiz Cerda JL, Gomez Perez L, Ramirez Backhaus M, Delgado Oliva F, Rebollo P, Gonzalez-Segura Alsina D, Arumi D; Grupo de Estudio Cooperativo EPICC. [Prevalence of urinary incontinence and hyperactive bladder in the Spanish population: results of the EPICC study]. Actas Urol Esp. 2009 Feb;33(2):159-66. doi: 10.1016/s0210-4806(09)74117-8. Spanish. PMID 19418840
- [Background] Rexach Cano, L., Verdejo Bravo, C. Incontinencia urinaria. Inf Ter Sist Nac Salud 1999; 23:149-159.
- [Background] Fantl JA, Newman DK, Colling J, DeLancey JO, Keeys C, Loughery R. Urinary Incontinence in Adults: Acute and Chronic Management Clinical Practice Guideline, N. 2, 1996 Update. AHCPR.
- [Background] Lyons SS, Specht JKP. Research-based protocol: prompted voiding for persons with urinary incontinence. The University of Iowa Gerontological Nursing Interventions Research Center, Research Development and Dissemination Core, 1999
- See also: Nursing Care Plan tool. NNNConsult. Elsevier; 2015. — http://www.nnnconsult.com/